CLINICAL TRIAL: NCT04325412
Title: Cardiac complicAtions in Patients With SARS Corona vIrus 2 regisTrY
Brief Title: Cardiac complicAtions in Patients With SARS Corona vIrus 2 (COVID-19) regisTrY
Acronym: CAPACITY-COVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Prof. Dr. F.W. Asselbergs, Prof. Dr. F.W. Asselbergs, UMC Utrecht
Other Study IDs: 20-161/C
Record Dates: First submitted 2020-03-25; First posted 2020-03-27 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: COVID-19; Cardiovascular Diseases
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CAPACITY (www.capacity-covid.eu) is a registry of patients with COVID-19 across Europe and has been established to answer questions on the role of cardiovascular disease in this pandemic. It is an extension of the Case Record Form (CRF) that was released by the ISARIC (International Severe Acute Respiratory and Emerging Infection Consortium) and WHO (World Health Organisation) in response to the emerging outbreak of COVID-19.

DETAILED DESCRIPTION:
The aim of CAPACITY is to collect data regarding the cardiovascular history, diagnostic information and occurrence of cardiovascular complications in COVID-19 patients. By collecting this information in a standardized manner, CAPACITY can aid in providing more insight in (1) the incidence of cardiovascular complications in patients with COVID-19, and (2) the vulnerability and clinical course of COVID-19 in patients with an underlying cardiovascular disease.

The CAPACITY extension to the ISARIC-WHO CRF consists of additional data collection instruments for:

* cardiac history and cardiovascular risk factors
* prior use of cardiac medication or NSAIDs
* electrocardiography (ECG)
* echocardiography
* cardiac MRI
* invasive cardiac procedures
* cardiac complications
* cardiac biomarkers
* cardiac outcome during admission

ELIGIBILITY:
Inclusion Criteria:

* Highly suspected/confirmed infection with SARS-CoV-2

Exclusion Criteria:

- Patients that opt-out

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients were admitted at one of the participating centres with highly suspected/confirmed infection with SARS-CoV-2.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2021-03-23 (Estimated); Study Completion 2021-06-23 (Estimated)

PRIMARY OUTCOMES:
The incidence of cardiovascular complications in patients with COVID-19 | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Henkens MTHM, Raafs AG, Verdonschot JAJ, Linschoten M, van Smeden M, Wang P, van der Hooft BHM, Tieleman R, Janssen MLF, Ter Bekke RMA, Hazebroek MR, van der Horst ICC, Asselbergs FW, Magdelijns FJH, Heymans SRB; CAPACITY-COVID collaborative consortium. Age is the main determinant of COVID-19 related in-hospital mortality with minimal impact of pre-existing comorbidities, a retrospective cohort study. BMC Geriatr. 2022 Mar 5;22(1):184. doi: 10.1186/s12877-021-02673-1. PMID 35247983
- See also: All study documents can be found on this website. — http://www.capacity-covid.eu